CLINICAL TRIAL: NCT04204941
Title: A Phase 1b/3 Global, Randomized, Double-blind, Placebo-Controlled Trial of Tazemetostat in Combination With Doxorubicin as Frontline Therapy for Advanced Epithelioid Sarcoma
Brief Title: Tazemetostat in Combination With Doxorubicin as Frontline Therapy for Advanced Epithelioid Sarcoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: FDA and Ipsen alignelment: Due to unfeasibility and the resulting inability to meet the required enrolment targets. No safety concerns
Sponsor: Epizyme, Inc. (Industry)
Responsible Party: Sponsor
Organization: Ipsen (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EZH-301; 2019-003648-55 (EudraCT Number)
Record Dates: First submitted 2019-12-11; First posted 2019-12-19 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Advanced Soft-tissue Sarcoma; Advanced Epithelioid Sarcoma
MeSH Terms: interventions — tazemetostat; Doxorubicin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Phase 1b: Open-label: Tazemetostat + Doxorubicin (Experimental): Phase 1b: On cycle 1 day -1, participants will receive a single morning dose of tazemetostat at the assigned dose level. Participants will receive doxorubicin 75 mg/m2 intravenously (IV) on day 1 of each cycle for up to 6 cycles.
  Tazemetostat will be escalated from a starting dose of 400 mg twice daily PO to 600 mg twice daily PO to 800 mg twice daily.
  Interventions: Drug: Tazemetostat; Drug: Doxorubicin HCl

INTERVENTIONS:
Drug: Tazemetostat — 400 mg, 600 to 800 mg of Tazemetostat will be administered twice daily.
  Other Names: EPZ-6438; IPN60200
Drug: Doxorubicin HCl — 75mg/m2 intravenous injection day 1 of each cycle for up to 6 cycles

SUMMARY:
The participants of this study will have advanced epithelioid sarcoma. Sarcoma is a cancer of the connective tissues, such as nerves, muscles and bones. Epithelioid sarcoma is an ultra-rare sarcoma of the soft-tissue.

Part 1 of this trial will evaluate the safety and the level of the study drug that the study drug combinations can be tolerated (known as tolerability). It is also designed to establish a recommended study drug dosage for the next part of the study.

Part 2 will evaluate and compare for each of the study drug combinations how long participants live without their disease getting worse.

The study drug is called tazemetostat. The study will test tazemetostat in combination with doxorubicin compared to placebo (dummy treatment) in combination with doxorubicin. Doxorubicin is a current front line treatment for epithelioid sarcoma

DETAILED DESCRIPTION:
The open-label phase 1b portion is designed to evaluate the safety of the combination of tazemetostat + doxorubicin, as well as to establish the maximum tolerated dose (MTD) and the Recommended Phase 3 Dose (RP3D). The phase 3 portion of the clinical trial aims to compare tazemetostat + doxorubicin to the current front-line standard treatment, single-agent doxorubicin + placebo, when used as first-line treatment in locally advanced unresectable or metastatic Epithelioid Sarcoma (ES).

The Phase 3 portion was planned but never initiated due to early termination during Phase 1b. Participants with confirmed Soft-tissue Sarcoma (STS) were enrolled in phases 1b.

ELIGIBILITY:
Inclusion Criteria

Participants must meet ALL the following inclusion criteria to be eligible to enroll in this study:

1. Have voluntarily agreed to provide written informed consent and demonstrated willingness and ability to comply with all aspects of the protocol. Study related activities will not start until written consent is obtained.
2. Life expectancy ≥ 3 months before enrollment
3. Phase 1b: 18-65 years old histologically confirmed Soft Tissue Sarcoma
4. Phase 3: ≥18 years old with unresectable locally advanced or metastatic Epithelioid Sarcoma and tumor tissue available
5. Have measurable disease
6. Eastern Cooperative Oncology Group Performance Status (ECOG) performance status of 0, 1, or 2
7. Have adequate hematologic (bone marrow (BM) and coagulation factors), renal and hepatic function as required per protocol
8. Females must not be lactating or pregnant at Screening or Baseline
9. Females must not be pregnant or breast feeding and agree to use highly effective contraception during the clinical trial and for 6 months following the final dose of study
10. Male participants of child-bearing potential must have had either a successful vasectomy or practice highly effective contraception
11. Participants diagnosed with human immunodeficiency virus (HIV) are eligible to participate in the study if their infection is well controlled on anti-retroviral therapy.

Exclusion Criteria

Participants meeting any of the following exclusion criteria are NOT eligible to enroll in this study:

1. Prior exposure to tazemetostat or other inhibitor(s) of enhancer of zeste homologue-2 (EZH2).
2. Prior systemic anticancer therapy.
3. Contraindications noted in the doxorubicin label
4. Have any prior history of myeloid malignancies, including myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML).
5. Have prior history of T-cell lymphoblastic lymphoma (T- LBL/)/T-cell acute lymphoblastic leukemia (T-ALL).
6. Have participated in another interventional clinical study and received investigational drug within 30 days or 5 half-lives, whichever is longer, prior to the planned first dose of study treatment.
7. Have known active central nervous system (CNS) or any leptomeningeal metastasis of primary extracranial tumor.
8. Participants taking medications that are known potent cytochrome P450 3A4 (CYP3A4) inducers/inhibitors (including St. John's Wort)
9. Are unwilling to exclude Seville oranges, grapefruit juice, AND grapefruit from the diet and all foods that contain those fruits from time of enrollment to through the duration of study participation.
10. Major surgery within 4 weeks before the first dose of study treatment. Participants must have recovered from surgery prior to enrollment to this study.
11. Are unable to take oral medication OR have malabsorption syndrome or any other uncontrolled gastrointestinal condition (eg, nausea, diarrhea, vomiting) that might impair the bioavailability of study treatment.
12. Have an active infection requiring systemic therapy.
13. Are immunocompromised (ie, has a congenital immunodeficiency).
14. Have known hypersensitivity to any component of tazemetostat or doxorubicin.
15. Cardiovascular impairment as stated in the protocol
16. Have a known active infection with hepatitis B virus (HBV, as measured by positive hepatitis B surface antigen), hepatitis C virus (HCV, as measured by positive hepatitis C antibody).
17. Any other major illness that, in the Investigator's judgment, will substantially increase the risk associated with the participant's participation in this study OR interfere with their ability to receive study treatment or complete the study.
18. Female participants who are pregnant or breastfeeding.
19. Participants who have undergone a solid organ transplant.
20. Participants with malignancies other than STS (phase 1b) or ES (Phase 3 only).
21. Participants housed in an institution by order of the authorities or courts.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-12-19 (Actual); Primary Completion 2024-06-14 (Actual); Study Completion 2024-06-14 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicities (DLTs) | 1 Cycle/21 days
  Determined by Adverse Events (AEs) and clinical laboratory tests.
Progression free survival (PFS) | Through study completion, an average of two years.
  Phase 3: Assessed by Independent Review Committee. Phase 3 was planned but never initiated; therefore, no data were collected for these endpoints

SECONDARY OUTCOMES:
Phase 1b: Pharmacokinetics (PK) of tazemetostat when administered in combination with doxorubicin in participants with soft tissue sarcoma (STS): Area under the Plasma Concentration Time Curve from time 0 to 24 hours (AUC0-24) | Cycles 1, 2, 3, and 5 of the first continuous 21-day cycles of combination therapy
Phase 1b: PK of tazemetostat when administered in combination with doxorubicin in participants with STS: Area under the Plasma Concentration Time Curve From time 0 to the last observable concentration (AUC0- last) | Cycles 1, 2, 3, and 5 of the first continuous 21-day cycles of combination therapy
Phase 1b: PK of tazemetostat when administered in combination with doxorubicin in Participants with STS: The maximum observed concentration (Cmax). | Cycles 1, 2, 3, and 5 of the first continuous 21-day cycles of combination therapy
Phase 3: Overall Survival (OS) | Through study completion, an average of two years.
  Phase 3 was planned but never initiated; therefore, no data were collected for these endpoints
Phase 3: Incidence of Adverse Events (AEs) | Through study completion, an average of two years.
  All AEs, including clinically significant laboratory parameters will be graded by the investigator according to the Common Terminology Criteria for Adverse Events (CTCAE). Phase 3 was planned but never initiated; therefore, no data were collected for these endpoints
Phase 3: PFS | Through study completion, an average of two years.
  Assessed by the investigator. Phase 3 was planned but never initiated; therefore, no data were collected for these endpoints
Disease control rate (DCR) | Through study completion, an average of two years
  Defined as the number of participants who achieve response complete response (CR) + partial response (PR) or who have stable disease (SD). Phase 3 was planned but never initiated; therefore, no data were collected for these endpoints.
Objective response rate (ORR) | Through study completion, an average of two years
  ORR is defined as the proportion of participants achieving complete or partial response. Determined based on the Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
Duration of treatment (DOR) | Through study completion, an average of two years
  Defined as the time from first documented evidence of CR or PR to the time of first documented disease progression or death, whichever occurs first
Change from baseline in European Organisation for Research and Treatment of Cancer (EORTC) Core Quality of Life Questionnaire (QLQC) (EORTC QLQC-30) | Through study completion, an average of two years
  The EORTC QLQC-30 physical function, role function, and global health status domains will be assessed
Progression-Free Survival on Next Line of Therapy (PFS2) | Through study completion, an average of two years
  Defined as time from randomization to objective tumor progression on next-line treatment or death, whichever occurs first
Time to first subsequent anti-cancer therapy ((TFST) | Through study completion, an average of two years
  Defined as the time from randomization to the time to first subsequent therapy
Population PK parameters of tazemetostat when administered in combination with doxorubicin: Oral clearance (CL/F) | Cycles 1, 2, 3, and 5 of the first continuous 21-day cycles of combination therapy
  CL/F is defined as the apparent oral clearance following administration of tazemetostat when administered in combination with doxorubicin
Population PK parameters of tazemetostat when administered in combination with doxorubicin: oral volume of distribution (Vss). | Cycles 1, 2, 3, and 5 of the first continuous 21-day cycles of combination therapy
Population PK parameters of tazemetostat when administered in combination with doxorubicin: Area Under the Curve at steady state (AUCss) | Cycles 1, 2, 3, and 5 of the first continuous 21-day cycles of combination therapy
Population PK parameters of tazemetostat when administered in combination with doxorubicin: trough concentration (Ctrough) | Cycles 1, 2, 3, and 5 of the first continuous 21-day cycles of combination therapy
Population PK parameters of tazemetostat when administered in combination with doxorubicin: Cmax | Cycles 1, 2, 3, and 5 of the first continuous 21-day cycles of combination therapy

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (21):
- United States (18):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Sarcoma Oncology Research Center, Santa Monica, California
  - University of Colorado Hospital - Anschutz Cancer Pavilion, Aurora, Colorado
  - Sarah Cannon Research Institute at HealthONE, Denver, Colorado
  - Mayo Clinic-Jacksonville, Jacksonville, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Insititute, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - Washington University, St Louis, Missouri
  - Columbia University Irving Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - The Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center - Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Sarah Cannon and HCA Research Institute, Nashville, Tennessee
  - Fred Hutchinson Research Center, Seattle, Washington
- McGill University Faculty of Medicine - Royal Victoria Hospital, Montreal, Quebec, Canada
- National Taiwan University Hospital, Taipei, Taiwan
- Royal Marsden Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, annotated case report form, statistical analysis plan, and dataset specifications.
  Patient level data will be anonymized and study documents will be redacted to protect the privacy of study participants.
Time Frame: Where applicable, data from eligible studies are available 6 months after the studied medicine and indication have been approved in the United States (US) and/or Europe (EU).
Access Criteria: Further details on Ipsen's sharing criteria and process for sharing are available here (https://www.ipsen.com/science/clinical-trials/clinical-data-transparency/).
URL: https://www.ipsen.com/science/clinical-trials/clinical-data-transparency/

REFERENCES:
- [Derived] Gounder M, Schoffski P, Jones RL, Agulnik M, Cote GM, Villalobos VM, Attia S, Chugh R, Chen TW, Jahan T, Loggers ET, Gupta A, Italiano A, Demetri GD, Ratan R, Davis LE, Mir O, Dileo P, Van Tine BA, Pressey JG, Lingaraj T, Rajarethinam A, Sierra L, Agarwal S, Stacchiotti S. Tazemetostat in advanced epithelioid sarcoma with loss of INI1/SMARCB1: an international, open-label, phase 2 basket study. Lancet Oncol. 2020 Nov;21(11):1423-1432. doi: 10.1016/S1470-2045(20)30451-4. Epub 2020 Oct 6. PMID 33035459